CLINICAL TRIAL: NCT03325920
Title: Validation of a Diagnostic Method for Quantification and Monitoring of Sleep Bruxism
Brief Title: Validation of a Diagnostic Method for Quantification of Sleep Bruxism
Acronym: DIABRUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017094440
Record Dates: First submitted 2017-09-22; First posted 2017-10-30 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Sleep Bruxism; Diagnosis
Keywords: sleep bruxism; diagnosis; validation study; assessment
MeSH Terms: conditions — Sleep Bruxism; Disease

STUDY DESIGN:
Intervention Model Description: Single-center, national, double-blind, controlled clinical trial with parallel group design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, as well as the investigating dentist are blind to the result obtained from the polysomnographic recording. The statistican is also unaware of the sleep bruxism diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep bruxism group (Experimental): 25 sleep bruxism subjects wear the DIABRUX for five consecutive nights.
  Interventions: Device: DIABRUX
- non-sleep bruxism group (Experimental): 25 non-sleep bruxism subjects wear the DIABRUX for five consecutive nights.
  Interventions: Device: DIABRUX

INTERVENTIONS:
Device: DIABRUX — All participants receive an individually fabricated diagnostic plate, viz the DIABRUX, for the upper or lower jaw to be worn for five consecutive nights. After use a newly developed analyzing software quantifies the abrasion on the diagnostic plate, thus resulting in a score, viz the Pixel score. This represents a quantitative measure of sleep bruxism activity.
  Other Names: Diagnostic plate

SUMMARY:
This study aims to validate a new diagnostic method for quantification and monitoring of sleep bruxism.

DETAILED DESCRIPTION:
Sleep bruxism has characteristically been defined by the American Academy of Sleep Medicine as 'an oral activity characterized by grinding or clenching of the teeth during sleep, usually associated with sleep arousals'. For sleep bruxism diagnosis, to date the polysomnographic recordings represent the highest standard for sleep bruxism diagnosis, but they are concomitantly associated with disadvantages which include technical complexity, limited availability, and the fact that they are time-consuming and cost-intensive. Recently, a prototype of a diagnostic plate has been developed which allows a fully-automatic, computer-based quantification of abrasion thereupon for the assessment of sleep bruxism activity. The results of the pilot study were promising, and therefore, the aim of the present study is to refine and validate this new diagnostic method for quantification and monitoring of sleep bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and understood the approved informed consent form and is able to meet the proposed study proceedings
* for the sleep bruxism Group: subjects have to fulfill the clinical criteria of the American Academy of Sleep Medicine (sleeping partner's Report of grinding sounds during sleep within the last 6 months, plus at least one of the following symptoms: abnormal attrition of the teeth or shiny spots on dental restorations, hypertrophy of the masseteric muscle upon palpation, and/or self-report of muscle fatigue on awakening. In addition to the clinical criteria for sleep bruxism diagnosis, the following polysomnographic criteria have to be present: bruxism episodes/hr >4, bruxism burst/hr >25, at least one episode of grinding per sleep period

Subjects that do not meet any of the clinical or polysomnographic criteria for sleep bruxism were included into the non-sleep bruxism group.

Exclusion Criteria:

* current participation in another interventional Investigation
* cardiac Pacemaker
* central nervous system and peripheral nervous system disorders
* use of sedating medications and/or psychopharmacologically effective drugs
* suspected severe psychological disorder (for example schizophrenia)
* a lack of German language
* drug and/or alcohol abuse
* pregnancy or breast-feeding

Participants of the sleep bruxism group that do not meet any of the clinical or polysomnographic criteria for sleep bruxism were excluded from the sleep bruxism group.

Participants of the non-sleep bruxism group that fulfill the clinical and/or polysomnographic criteria for sleep bruxism were excluded from the non-sleep bruxism group.

Further dental exclusion criteria are:

* prostheses or extensive prosthetic restorations
* dental functional treatment during the last 6 months
* gross malocclusion
* too many missing teeth that omit fabricating a diagnostic plate
* fixed brace
* temporomandibular dysfunction requiring treatment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Pixel score of the diagnostic plate | The DIABRUX plate should be worn for five consecutive nights. This will be performed by each participant at the earliest of the 12th and not later than the 85th days after screening.
  Quantitative measure of sleep bruxism activity

SECONDARY OUTCOMES:
Psychologic load | Subjects who fulfill the inclusion criteria and none of the exclusion criteria should stipulate the first visit not later than 28 days after screening (day 0).
  Psychologic load will be estimated by means of the Symptom-Check-List-90 Standard (SCL-90-S; Franke, 1995) measuring subjective complaints, as well as physical and mental impairments. This self-assessment questionnaire implies 90 items with a total of 9 different scales: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism and seven supplementary questions. Every item starts with "For the past week, how much were you bothered by" followed by 90 different symptoms. The items are Likert scaled with a range from 0 ("not at all") to 4 ("extremely"), whereby higher values represent a higher psychological load. Three global indices are reported via the SCL-90-S, viz. the Global Severity Index (GSI), the Positive Symptom Total (PST), and the Positive Symptom Distress Index (PSDI). The higher the score of each index, the greater is the psychological load.
Oral health-related quality of life | Recorded during the 1. visit; this appointment may happen between the 1st-28th day of study participation.
  Oral health-related quality of life will be recorded with the Oral Health Impact Profile German 14 (OHIP-G14; Slade, 1997). The OHIP-G14 measures the subjective experience in terms of oral health (teeth, mouth, jaw and denture). It contains 14 questions (e.g. "Have you had painful aching in your mouth?") which are Likert scaled from 0 ("never") to 4 ("very often"). All questions refer to the last month. There are 7 different dimensions with two questions each (functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap). Values can be summed up to a total score, ranging between 0 and 56. Higher scores represent a more negative experience with one's oral health.
Pain perception | Recorded during the 1. visit; this appointment may happen between the 1st-28th day of study participation.
  Pain perception will be calculated using the pain perception scale (Schmerzempfindungsskala, SES; Geissner, 1996). The SES is a self-assessment questionnaire for describing the subjective pain perception. It consists of two parts (part A with 14 items and part B with 10 item) which form two global scales: A = affective pain perception and B = sensoric pain perception. Every single item is based on adjective sentences like "I feel my pain is burning". Items are Likert scaled with a range from 1 ("this is not true") to 4 ("this is exactly true"). Higher values correspond to a painfully experience and represent a worse outcome. Item values are summed for every scale, therefore the scale range A is from 14 to 56 and the scale range B is from 10 to 40. Raw scale values can be transferred into the percent range.
Dream experience | Recorded during the 2. and the 3. visit; this appointment may happen between the 2nd-57th day of study participation.
  Aspects of dream experience will be assessed using the Mannheim Dream Questionnaire (MADRE; Schredl et al., 2014) combined with a dream protocol. These include dream recall, dream types, attitude towards dreaming, what dreamers do with their dreams, and effects of dreaming on waking life. Every item measures a single aspect of dreaming and the response format gathers information about frequencies (e.g. "every morning" or "less than once a month") and contents (e.g. topics of nightmares in childhood). Scaling of the items varies between 3 to 8 points and they range between 0 (least degree of manifestation/frequency) and maximum 8 (highest degree of manifestation/frequency). No global score exists. There is one aggregate score concerning attitude towards dreams, that encompasses 6 items with a 5-point Likert scale (0 = "not at all" to 4 "totally"), e.g. "I think that dreaming is in general a very interesting phenomenon."
Individual stress coping | Recorded during the 4. visit; this appointment may happen between the 5th-71th day of study participation.
  The stress coping questionnaire 78 (SVF-78; Janke et al., 1985) assesses individual long-term and constant strategies to cope with stress. The respondents determine by themselves how likely they apply 78 different coping styles. Coping styles refer to everyday situations. Every items starts with the phrase "If I was affected, disturbed or unsettled by someone or something", followed by a coping strategy (e.g. "I ask someone to help me"). Items are Likert scaled with a range from 0 ("not at all") to 4 ("very likely"). Higher values stand for a higher likelihood to apply the reaction in a certain situation. Two different main scales exist which sum up either positive strategies (adaptive strategies) or negative strategies (maladaptive strategies). Higher scores in positive strategies represent a stress reductive coping style. Higher scores in negative strategies represent a stress enhancing coping style. Raw values can be transferred to standardized T-scores.
State-trait-Anxiety | Recorded during the 4. visit; this appointment may happen between the 5th-71th day of study participation.
  The State-Trait-Anxiety Inventory (STAI; Laux et al. 1981) consists of 2 questionnaires with 20 items, respectively, and provides 20 different statements to describe ones feelings of anxiety at the moment. Half of the statements contain anxiety-present (e.g. "I feel over-excited and rattled"), the other half anxiety-absent items (e.g. "I am relaxed"). 4-point Likert scales are used with values from 1 ("not at all") to 4 ("very much so"). The trait anxiety scale comprises 20 statements to describe feelings of anxiety in general. 13 statements involve anxiety-present (e.g. "I lack self-confidence") and 7 anxiety-absent items (e.g. "I feel secure"). 4-point Likert scales allow data indication with values from 1 ("almost never") to 4 ("almost always"). The range of values is between 20 and 40 for each scale. The higher the score the more intense is the feeling of anxiety or, in relation to trait anxiety, the heavier is the anxiety disorder.
Subjective rating of the DIABRUX characteristics | The short questionnaire should be returned to the site together with the used DIABRUX plate. This will be performed by each participant at the earliest of the 12th and not later than the 85th days after screening.
  Subjective rating of the device characteristics will be evaluated by using a short questionnaire.

OTHER OUTCOMES:
Assessment of probable sleep bruxism (clinical AASM criteria) | Recorded during the 1. visit; this appointment may happen between the 1st-28th day of study participation.
  Probable sleep bruxism will be estimated by combining self-report plus the inspection part of a clinical dental examination according to the clinicial AASM criteria (AASM, 2005).
Assessment of probable awake bruxism | Recorded during the 1. visit; this appointment may happen between the 1st-28th day of study participation.
  Awake bruxism (diurnal clenching) will be measured on the basis of self-report plus the inspection part of a clinical examination.
Presence of different forms of temporomandibular disorders | Recorded during the 1. visit; this appointment may happen between the 1st-28th day of study participation.
  The presence of different forms of temporomandibular disorders will be verified by means of the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Ommerborn, Dr., Principal Investigator — Universitätsklinikum Düsseldorf/Heinrich-Heine-University Düsseldorf
Locations (1):
- Poliklinik für Zahnerhaltung, Parodontologie und Endodontologie Universitätsklinikum der Heinrich-Heine- Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ommerborn MA, Giraki M, Schneider C, Schaefer R, Gotter A, Franz M, Raab WH. A new analyzing method for quantification of abrasion on the Bruxcore device for sleep bruxism diagnosis. J Orofac Pain. 2005 Summer;19(3):232-8. PMID 16106717